CLINICAL TRIAL: NCT06710899
Title: Does Vitamin C Improve the Efficacy of Methenamine Hippurate (Hiprex®) in Prophylaxis of Recurrent Urinary Tract Infections? A Proof of Concept Study
Brief Title: Vitamin C and Hiprex in rUTI
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3399
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — methenamine hippurate; Ascorbic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment phase A (Experimental): Methenamine Hippurate 1g BD for 6 months
  Interventions: Drug: Methenamine Hippurate 1g BD
- Treatment phase B (Experimental): Methenamine Hippurate 1g BD + Vitamin C 1g BD for 6 months
  Interventions: Drug: Methenamine Hippurate 1g BD + Vitamin C 1g BD
- Treatment phase C (Experimental): Methenamine 1g BD for 6 months
  Interventions: Drug: Methenamine Hippurate 1g BD

INTERVENTIONS:
Drug: Methenamine Hippurate 1g BD — Methenamine Hippurate 1g BD for 6 months
  Arms: Treatment phase A; Treatment phase C
Drug: Methenamine Hippurate 1g BD + Vitamin C 1g BD — Methenamine Hippurate 1g BD + Vitamin C 1g BD for 6 months
  Arms: Treatment phase B

SUMMARY:
A single centre proof of concept study to assess whether Vitamin C improves the efficacy of Methenamine Hippurate (Hiprex®) in the prophylaxis of recurrent urinary tract infections (rUTIs) in women

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥18 years
* Recurrent proven UTI, defined as "two or more proven infections in six months or three or more infections in six months"
* Willing and able to give fully informed consent
* Patients suitable for prophylaxis following discussion with their clinician.
* No contra-indications to treatment with methenamine hippurate or Vitamin C
* All women will have undergone standard diagnostic work-up and have followed routine conservative UTI prevention measures.
* A working email address to be used to submit urine pH results
* Willing and able to comply with the study procedures
* Females of childbearing potential must be willing to use a highly effective method of contraception (hormonal or barrier method of birth control; abstinence; sterilisation or vasectomised partner)

Exclusion Criteria:

* Males
* Women who are pregnant or breast-feeding
* Contraindications to methenamine hippurate as described in BNF: known allergy, gout, severe metabolic acidosis, severe dehydration, eGFR less than 10 ml/min, severe hepatic impairment
* Currently using vitamin C containing supplement or cranberry extract tablets
* Women using urinary alkalinisation agents, e.g potassium citrate, sodium bicarbonate
* Currently receiving any form of bladder instillation or intradetrusor Onabotulinum Toxin A injections
* Patients already on low-dose antibiotics or methenamine hippurate (due to delay that will be incurred by 3-month washout period)
* Indwelling urinary catheter in situ or performing clean intermittent self-catheterisation
* Correctable urinary tract abnormalities, e.g., urinary tract calculi, urinary retention
* Formation of ileal conduit or augmented bladder
* Neurogenic bladder dysfunction
* Hyperoxaluria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of UTIs | 24 months
  The incidence of symptomatic UTI during each six-month treatment phase of either methenamine hippurate alone or methenamine hippurate plus vitamin C

SECONDARY OUTCOMES:
Urine pH | 24 months
  Measurement of urine pH during each treatment phase

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire, United Kingdom